CLINICAL TRIAL: NCT03297424
Title: A Phase 1b Dose-escalation Study to Assess Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PLX2853 in Subjects With Advanced Malignancies
Brief Title: A Study of PLX2853 in Advanced Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opna Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX124-01
Record Dates: First submitted 2017-09-08; First posted 2017-09-29 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Small Cell Lung Cancer; Uveal Melanoma; Ovarian Clear Cell Carcinoma; Non-Hodgkin Lymphoma; Advanced Malignancies; Solid Tumor; Diffuse Large B Cell Lymphoma; Follicular Lymphoma
Keywords: PLX2853; Small cell lung cancer (SCLC); Uveal Melanoma; Ovarian Clear Cell Carcinoma; Non-Hodgkin Lymphoma; Advanced Malignancies; Solid Tumor; Diffuse Large B Cell Lymphoma (DLBCL); Follicular Lymphoma (FL); ARID1A
MeSH Terms: conditions — Small Cell Lung Carcinoma; Uveal Melanoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLX2853 (Experimental): Phase 1b (Dose Escalation): Approximately 45 subjects with advanced malignancies to establish the MTD/RP2D. Up to 6 additional subjects may be enrolled at the MTD/RP2D as a dose confirmation.
  Phase 2a (Dose Expansion): There will be 5 total expansion cohorts. Either 10 or 29 subjects per cohort in each of 4 expansion cohorts: advanced SCLC, uveal melanoma, OCCC, and any other advanced malignancy with a known ARID1A mutation (between 40 to 116 subjects total for the solid tumor expansion phase). For the 5th expansion cohort, up to 20 subjects may be enrolled for NHL.
  Interventions: Drug: PLX2853

INTERVENTIONS:
Drug: PLX2853 — tablets
  Other Names: PLX2853 tablets

SUMMARY:
The purpose of this research study is to evaluate safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of the investigational drug PLX2853 in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of the following:
* Phase 1b:

  * Histologically confirmed advanced refractory solid tumor that is measurable or evaluable per RECIST 1.1 criteria.
  * Histologically confirmed NHL: diffuse large B-cell lymphoma and follicular lymphoma (Grade 1-3A) which is measurable or evaluable per Lugano criteria, has progressed following at least 1 line of prior anticancer therapy.
* Phase 2a: Patients with various solid tumors or NHL who have received prior therapy.
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Adequate organ function as appropriate for the disease under study. All screening laboratory tests should be performed within 10 days of treatment initiation.
* Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test at Screening (≤7 days prior to 1st study drug dose) and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 90 days after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year.
* Fertile men must agree to use an effective method of birth control during the study and for up to 90 days after the last dose of study drug.
* All associated clinically significant drug-related toxicity from previous cancer therapy must be resolved prior to study treatment administration (alopecia, erectile impotence, hot flashes, decreased libido, and neuropathy is allowed).
* Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements

Exclusion Criteria:

* Prior exposure to a bromodomain inhibitor, such as OTX-015 or CPI-0610
* Known uncontrolled fungal, bacterial, and/or viral infection ≥Grade 2
* Autoimmune hemolytic anemia or autoimmune thrombocytopenia
* Presence of symptomatic or uncontrolled central nervous system or leptomeningeal metastases
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Clinically significant cardiac disease such as cardiac arrhythmias including bradyarrhythmias and/or subjects who require anti-arrhythmic therapy (excluding beta blockers or digoxin), including uncontrolled hypertension or arterial or venous thrombotic events. Subjects with controlled atrial fibrillation are not excluded.
* Inability to take oral medication or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption
* Non-healing wound, ulcer, or bone fracture
* Subject has known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection or is known to be a carrier of hepatitis B or C. Subjects who are positive for hepatitis C virus (HCV) antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible. Subjects with occult or prior hepatitis B virus (HBV) infection (defined as positive total hepatitis B core antibody (HBcAb) and negative hepatitis B surface antigen (HBsAg) may be included if HBV DNA is undetectable. These subjects must be willing to undergo additional testing per local standard of care.
* Active second malignancy with the exception of any of the following:

  * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer;
  * Adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for ≥2 years;
  * Low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 ng/mL; or
  * Any other cancer from which the patient has been disease-free for ≥3 years.
* Subjects with documented hepatic metastases involving >50% of the hepatic parenchyma, or any individual liver metastasis >5 cm, as assessed by the investigator.
* Major surgery or significant traumatic injury within 14 days prior to Cycle 1 Day 1
* Receipt of anti-cancer therapy with insufficient washout prior to Cycle 1 Day 1: No chemotherapy, radiation therapy, or small molecule tyrosine kinase inhibitors (TKI) for the treatment of cancer within 14 days or 5 half-lives (whichever is shorter) of Cycle 1 Day 1. Certain standard of care hormonal anticancer therapies, such as agents targeted to GnRH for the treatment of prostate cancer or aromatase inhibitors for the treatment of breast cancer, may be permitted after consultation with the medical monitor. No immune therapy or other biologic therapy (other monoclonal antibodies or antibody-drug conjugates [ADCs]) for the treatment of cancer within 28 days of Cycle 1 Day 1.
* Subject is receiving systemic steroids at doses greater than the equivalent of prednisone 10 mg daily, with the exception of intermittent use for the treatment of emesis
* Subject is participating in any other therapeutic clinical study (observational or registry trials are allowed)
* Female subjects who are pregnant or breast-feeding
* Presence of any other medical, psychological, familial, sociological, or geographic condition potentially hampering compliance with the study protocol or would interfere with the study endpoints or the subject's ability to participate in the study in the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | First dose of study drug through at least 30 days after end of treatment.
Area under the concentration-time curve (AUC) of PLX2853. | From first dose of PLX2853 up to 30 days after end of treatment.
Maximum observed concentration (Cmax) of PLX2853. | From first dose of PLX2853 up to 30 days after end of treatment.
Time to peak concentration (Tmax) of PLX2853. | From first dose of PLX2853 up to 30 days after end of treatment.
Half life (t1/2) of PLX2853. | From first dose of PLX2853 up to 30 days after end of treatment.
Number of participants who experience dose limiting toxicity as defined in the protocol. | Up to 2 years
  The highest dose level at which less than 2 of 6 participants or less than 33% of participants (if cohort is expanded beyond 6) experience a dose limiting toxicity will be considered the maximum tolerated dose / recommended phase 2 dose.
Change in disease burden using RECIST 1.1 (solid tumors) or Lugano criteria (NHL). | Up to 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) defined according to standard criteria for the relevant malignancy [Phase1b] | From the first dose of study drug until the date of documented response to treatment, assessed up to 2 years.
Duration of response (DOR) | DOR defined as the time from the initial objective response to disease progression or death, whichever occurs first, assessed up to 2 years.
Progression-Free Survival (PFS) | PFS time is defined as the time from the first dose of PLX2853 to disease progression or death, whichever occurs first, assessed up to 2 years.
Overall Survival (OS) | From the first dose of study drug until the date of death from any cause, assessed up to 2 years.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Honor Health, Scottsdale, Arizona
  - Sylvester Comprehensive Cancer Center / University of Miami Miller School of Medicine, Miami, Florida
  - Columbia University Medical Center, New York, New York
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia